CLINICAL TRIAL: NCT02056080
Title: Observational, Retrospective and Multicenter Study to Evaluate the Clinical Benefit of Trastuzumab in Combination With Lapatinib in Metastatic Breast Cancer HER2 Positive Patients Who Has Been Previously Treated With Trastuzumab and/or Lapatinib
Brief Title: Clinical Benefit of the Treatment With Trastuzumab in Combination With Lapatinib in Metastatic Breast Cancer HER2 Positive Patients Who Has Been Previously Treated With Trastuzumab and/or Lapatinib
Acronym: TRASTYVERE
Status: Completed | Type: Observational
Sponsor: MedSIR (Other)
Responsible Party: Sponsor
Other Study IDs: MED-DBL-2012-01
Record Dates: First submitted 2014-01-10; First posted 2014-02-05 (Estimated); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Breast Neoplasm
Keywords: Breast Neoplasm; Receptor,HER2; Antineoplastic agent; Antibodies, monoclonal; Trastuzumab, Lapatinib; Protein kinase inhibitors; quinazolines
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A retrospective, observational, not EPA, multicenter study to evaluate the Clinical Benefit of Trastuzumab in Combination With Lapatinib in Metastatic Breast Cancer HER2 Positive Patients Who Has Been Previously Treated With Trastuzumab and/or Lapatinib between January 2005 and December 2011

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of metastatic breast cancer HER2-positive phenotype (confirmed by IHC 3 + or FISH positive)
* Older than 18 years
* Progressed to at least one prior treatment line for MBC with trastuzumab and / or lapatinib, either as monotherapy or in combination with chemotherapy or hormonal therapy schemes
* Having the patient's complete medical history that contains all lines antiHER2 therapy treatment
* Being a patient who initiated the combination of trastuzumab and lapatinib between January 2005 and December 2011
* Inform the patient and get the signature of the informed consent

Exclusion Criteria:

* Not having phenotypic classification of the tumor by IHC or FISH test for HER2
* Being a patient with HER2-negative phenotype(FISH negative or IHC in range [0-2 +] without FISH)
* Being a patient who received the trastuzumab and/or lapatinib treatment (TL) in combination with chemotherapy
* Being a patient who, since January 2012, began TL therapy for metastatic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HER2 positive metastatic breast cancer who progressed to antiHER2 therapy with trastuzumab and / or lapatinib for the metastasic disease and that between January 2005 and December 2011, began treatment with the combination of trastuzumab and lapatinib (TL).
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Clinical response rate assessed by RECIST criteria | Up to 24 weeks from the first clinical response rate assessment
  clinical benefit rate (CBR): defined as the percentage of patients who achieved an objective response (CR or PR) or tumor stabilization for at least 24 weeks or more during the period of treatment with the combination TL.
  This variable will be assessed by RECIST v 1.1

SECONDARY OUTCOMES:
To evaluate the progression-free survival in patients treated TL combination , previously treated with trastuzumab and / or lapatinib | Up to one year from the last dose of TL
  The progression will be evaluated by RECIST v 1.1.
To compare the clinical benefit and time to intra-patient progression between the combination TL and previous treatment lines. | Up to 24 weeks from the last dose of TL
  clinical benefit: defined as reaching a (complete or partial) objective response or stabilization of tumor for more than 24 weeks
To compare the time to progression of different subpopulations according to the biological characteristics of the tumor. | Up to one year from the last dose of TL
  The progression will be evaluated by RECIST v 1.1.
To identify the toxicity profile of the combination TL as a factor related to the intra-patient clinical benefit | Up to one year from the last dose of TL
  Adverse reactions observed during treatment of the combination TL, measured with scale CTCAE v.4

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin Gávila, MD, Principal Investigator — Valencia
Locations (11):
- Spain (11):
  - Barcelona
  - Córdoba
  - Girona
  - Jaén
  - Madrid
  - Pamplona
  - Salamanca
  - Santiago de Compostela
  - Seville
  - Valencia
  - Zaragoza